CLINICAL TRIAL: NCT05037786
Title: Exploring the Effect of a Brief Pain Education Intervention on Elite Athletes: Randomized Pilot Trial
Brief Title: Effects of Pain Neuroscience Education Using an Infographic in Basketball Elite Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaga (Other)
Responsible Party: Principal Investigator, Alejandro Luque-Suarez, Senior Lecturer, University of Malaga
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Infographic in elite athletes
Record Dates: First submitted 2021-08-31; First posted 2021-09-08 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Elite Basketball Athletes

STUDY DESIGN:
Intervention Model Description: In the control group, there will be a face-to-face intervention of 15 minutes of education on pain explained by Verbal form with supporting Powerpoint presentation. In the intervention group, the same pain education will be carried out, explained verbally but with the support of an infographic instead of a Powerpoint. The educational intervention will be carried out by one of the Unicaja Baloncesto Physiotherapists (research assistant), previously instructed by the research team.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Powerpoint group (Active Comparator): In the control group, there will be a face-to-face intervention of 15 minutes of education on pain explained by Verbal form with supporting Powerpoint presentation. The educational intervention will be carried out by one of the Unicaja Baloncesto Physiotherapists (research assistant), previously instructed by the research team.
  Interventions: Behavioral: Powerpoint
- Infographic group (Experimental): In the intervention group, the same pain education will be carried out, explained verbally but with the support of an infographic instead of a Powerpoint. The educational intervention will be carried out by one of the Unicaja Baloncesto Physiotherapists (research assistant), previously instructed by the research team.
  Interventions: Behavioral: Infographic

INTERVENTIONS:
Behavioral: Infographic — Key themes related to pain and injury in elite players based on previous studies presented using an A3 infographic
  Arms: Infographic group
Behavioral: Powerpoint — Key themes related to pain and injury in elite players based on previous studies presented using a Powerpoint
  Arms: Powerpoint group

SUMMARY:
The objective of this study is to analyze the effectiveness of a brief educational intervention supported by an infographic versus that supported by PowerPoint on the understanding of pain in elite athletes.

Secondary objective: to analyze whether a greater understanding of pain has effects on the intensity, extent and characteristics of pain experienced in the year after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Elite athletes over 18 years of age from the ACB Unicaja Basketball team during years 2021-2022

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2022-01-15 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
intensity, extent and characteristics of pain | 1 year follow up
  PainDETECT questionnaire (self-reported)

SECONDARY OUTCOMES:
Understanding of pain | baseline and immediately after the intervention
  Pain Neurophysiology Questionnaire (self-reported)

OTHER OUTCOMES:
Sociodemographic variables (age, gender, country of origin, height, weight) | baseline
  single questions

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Luque-Suarez, Study Director — University of Malaga
Locations (1):
- Mar Flores Cortes, Málaga, Spain

IPD SHARING:
Plan to Share IPD: No